CLINICAL TRIAL: NCT01706523
Title: An Open-Label Extension Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of STX209 (Arbaclofen) in Subjects With Autism Spectrum Disorders
Brief Title: Open Label Extension Study of STX209 (Arbaclofen) in Autism Spectrum Disorders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209AS209
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Autism; Asperger; Pervasive Developmental Disorder - Not otherwise specified
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STX209 (Experimental): Active treatment with STX209
  Interventions: Drug: STX209 (arbaclofen)

INTERVENTIONS:
Drug: STX209 (arbaclofen) — Long-term, daily, orally-administered STX209

SUMMARY:
This is an open-label extension protocol that will provide necessary data on the safety, tolerability, pharmacokinetics and efficacy of STX209 among subjects with ASD.

DETAILED DESCRIPTION:
This is an open label extension study enrolling by invitation only to those subjects that have completed Seaside protocols 209AS208 and 22007.

Protocol 209AS208, "A Randomized,Double-Blind, Placebo-Controlled, Study of the Efficacy, Safety, and Tolerability of STX209 (Arbaclofen) Administered for the Treatment of Social Withdrawal in Subjects with Autism Spectrum Disorders."

Protocol 22007, "An Open Label Extension Study to Evaluate the Safety, Tolerability and Pharmacokinetics of STX209 in Subjects with Autism Spectrum Disorder."

This open-label extension will provide data on the following:

1. Evaluate the safety and tolerability of long term use of STX209 (Arbaclofen)
2. Provide supporting pharmacokinetic analyses
3. Assess long term efficacy on social behaviors in subjects with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed study 22007 or 209AS208, and showed he can adequately follow the protocol, and with adequate medical justification to enter this study.
* Parent or other legally-authorized representative or caregiver is willing and able to perform all protocol-specified functions.
* Treatment with no more than 2 psychoactive medications
* Subjects with a history of seizure disorder must be adequately well-controlled, as specified in the study protocol
* For female subjects, negative pregnancy test

Exclusion Criteria:

* Comorbid conditions that might interfere with the conduct of the study or confound the interpretation of the study data, or endanger the subject.
* Current use of illicit drugs or alcohol abuse.
* Subjects with a serious adverse event or other adverse event in study 22007 or 209AS208 that was related to STX209, and that endangers the subject, in the opinion of the investigator
* Current use of another investigational drug, or of vigabatrin, tiagabine, or riluzole

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of STX209 | 100 weeks
  Spontaneously-reported adverse events, physical examination, and clinical laboratory assessments

SECONDARY OUTCOMES:
Aberrant Behavior Checklist | 100 weeks
  Open-label assessment of change from baseline on the ABC

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, M.D., Study Director — Seaside Therapeutics, Inc.
Locations (25):
- United States (25):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - UCDavis M.I.N.D Insitute, Sacramento, California
  - Pharmax Research Clinic, Miami, Florida
  - Lake Mary Pediatrics, Orange City, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Institute for Juvenile Research, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Missouri, Thompson Research Center for Autism & Neurodevelopmental Disorders, Columbia, Missouri
  - Seaver Autism Center, Mount Sinai Medical Center, New York, New York
  - NYS Institute for Basic Research in Developmental Disabilities, Staten Island, New York
  - UNC Chapel Hill Department of Psychiatry, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee Medical Group, LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, P.A., Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington